CLINICAL TRIAL: NCT05942508
Title: An Open, Single Arm, Single Center Phase Ib Clinical Trial to Evaluate the Efficacy and Safety of TQB2450 Combined With Anlotinib as Maintenance Therapy in Patients With Limited Stage Small Cell Lung Cancer Without Progression After First-line Radiotherapy and Chemotherapy
Brief Title: A Phase Ib Study of TQB2450 Combined With Anlotinib in Patients With Limited Stage Small Cell Lung Cancer After First-line Radiotherapy and Chemotherapy
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jinming Yu (Other)
Responsible Party: Sponsor-Investigator, Jinming Yu, Principal investigator, Shandong Cancer Hospital and Institute
Organization: Shandong Cancer Hospital and Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB2450-ALTN-Ib-02
Record Dates: First submitted 2023-06-07; First posted 2023-07-12 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Limited Stage Small Cell Lung Cancer; Not Progressed After First-line Chemoradiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB2450 Injection + Anlotinib Hydrochloride Capsules (Experimental): TQB2450 injection: 1200 mg/time, intravenous drip, day 1, Q3W; Anlotinib Hydrochloride Capsules: 8 mg/dose, once daily (QD), continuously used for 2 weeks, stopped for 1 week, and taken orally before breakfast (the starting dose of Anlotinib Hydrochloride is 8 mg, and it is allowed to be increased to 10 mg after two cycles of use)
  Interventions: Drug: TQB2450 Injection + Anlotinib Hydrochloride Capsules

INTERVENTIONS:
Drug: TQB2450 Injection + Anlotinib Hydrochloride Capsules — Anlotinib Hydrochloride Capsules: multi-target receptor tyrosine kinase inhibitor; TQB2450 injection: programmed cell death protein 1 (PD-1) human monoclonal antibody

SUMMARY:
To assess the efficacy and safety of TQB2450 in combination with anlotinib as maintenance therapy in patients with limited-stage small cell lung cancer who do not progress after first-line chemoradiotherapy. Based on the incidence and severity of benign and serious adverse events, as well as abnormal laboratory

ELIGIBILITY:
Inclusion Criteria:

* The subject voluntarily joins the study, signs the informed consent form, and has good compliance;
* Age: 18~75 years old (when signing the informed consent form); ECOG PS score: 0-1 points; Expected survival beyond 6 months; body weight> 40 kg;
* Patients with pathologically confirmed limited-stage small cell lung cancer (according to the Veterans Administration Lung Study Group (VALG stage);
* Through the neck, chest, abdomen, pelvic enhanced CT and brain plain scan + enhanced MRI examination with diagnostic quality, there is no evidence of metastatic disease (PET-CT examination is recommended before starting radiotherapy and chemotherapy, if not performed before radiotherapy and chemotherapy PET-CT examination, bone scan examination should be performed; PET-CT examination must be performed during the screening period after chemoradiotherapy to exclude metastasis);
* It is expected that no tumor resection will be required during the study (patients who are not suitable for surgery or those who are unwilling to undergo surgery are acceptable);
* Radiotherapy technology adopts three-dimensional conformal radiotherapy, conformal intensity-modulated radiotherapy, tomographic radiation therapy and other precision radiotherapy technologies;
* Patients must achieve CR, PR or SD after receiving radical platinum-based CRT and cannot develop disease progression;
* Patients with at least one measurable lesion confirmed according to RECIST 1.1 criteria prior to chemoradiotherapy;

Exclusion Criteria:

* Complex small cell lung cancer confirmed by histopathology or cytopathology;
* Subjects with known central nervous system metastasis and/or cancerous meningitis;
* Malignant pleural effusion and pericardial effusion;
* Imaging shows that the tumor has invaded important blood vessels, or the researcher has determined that the tumor is highly likely to invade important blood vessels and cause fatal massive bleeding during subsequent studies;
* Within 2 weeks before the start of the study treatment, he has received the treatment of traditional Chinese patent medicines and simple preparations with anti-tumor indications specified in the NMPA approved drug manual;
* Patients who have received immunomodulatory drugs within 30 days before starting treatment;
* Previously received anti PD-1, anti PD-L1, or anti PD-L2 drugs or medication targeting another stimulating or co inhibitory T cell receptor;
* Previous use of antivascular survival drugs（ bevacizumab, arotinib, apatinib ,ect);

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-05-30 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Adverse event | Start from the first dose until the last dose to within 84 days after the last dose or start new target indication treatment (whichever occurs first)
  Incidence and severity of adverse events
serious adverse event | Start from the first dose until the last dose to within 84 days after the last dose or start new target indication treatment (whichever occurs first)
  Incidence and Severity of Serious Adverse Events

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to approximately 36 months
  ORR:According to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.the proportion of subjects whose tumors are evaluated as complete response(CR) and partial response(PR) by subcenter imaging evaluation. It is recorded from the first use of the drug to disease progression or initiation of a new anticancer treatment.
disease control rate | Up to approximately 36 months
  The percentage of patients who have achieved remission or stable changes in their condition after treatment compared to the evaluable cases
duration of remission | Up to approximately 36 months
  The time from the first assessment of the tumor as CR or PR to the first assessment as PD (Progressive Disease) or death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital Affiliated to Shandong First Medical University, Jinan, Shandong, China

REFERENCES:
- [Derived] Liu X, Yin X, Zhuang L, Wen J, Wei Z, Cui W, Yu M, Zhao K, Liu L, Kong L, Jiang L, Jing X, Zhu H, Wang X, Dong X, Yu J, Meng X. Efficacy and safety of TQB2450 combined with anlotinib as maintenance therapy for LS-SCLC after definitive concurrent or sequential chemoradiotherapy: a prospective phase Ib study. BMC Cancer. 2025 Mar 20;25(1):509. doi: 10.1186/s12885-025-13885-8. PMID 40114144